CLINICAL TRIAL: NCT00004576
Title: AMPA Receptor Blockade With LY300164 in the Treatment of Parkinson's Disease
Brief Title: Study of LY300164 for the Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000084; 00-N-0084
Record Dates: First submitted 2000-02-17; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Dyskinesias; Parkinson Disease
Keywords: Dyskinesias; Glutamate; Levodopa; Parkinson's Disease
MeSH Terms: conditions — Dyskinesias; Parkinson Disease | interventions — talampanel

INTERVENTIONS:
Drug: LY300164

SUMMARY:
This study will test the effectiveness of an experimental drug called LY300164 on improving Parkinson's disease symptoms, such as movement impairments and tremor, as well as involuntary movements produced by long-term treatment with levodopa.

Patients with relatively advanced (Stage II to IV) Parkinson's disease between 30 and 75 years of age may be eligible for this 8-week study. Participants will have a complete medical history and physical examination, including blood tests and an electrocardiogram, and possibly brain magnetic resonance imaging (MRI), CT scan, and chest X-ray.

Patients will stop taking all anti-parkinsonism medications except levodopa (Sinemet) and the experimental drug during the study. For the first 1 to 3 days, patients will be in the hospital for a levodopa "dose-finding" procedure. For this study, levodopa is infused through a vein for up to 8 hours, with symptoms monitored frequently to determine the doses that will produce two results: 1) the dose that is less than what is needed to relieve symptoms, and 2) the dose that relieves symptoms, but may produce dyskinesias.

When these dose rates are determined, patients will begin treatment in one of two groups. One will take LY300164 3 times a day, along with levodopa, for 3 weeks. The second group will take placebo tablets (a look-alike tablet with no active ingredient) and levodopa on the same schedule as the LY300164 group. A brief medical examination and routine blood and urine tests will be done weekly. The drug dose will be increased every 3 to 4 days until significant side effects occur or the maximal dose is reached. Patients will be closely monitored for 4 hours after every increase. At the end of the 3 weeks, or when the maximal dose is reached, patients will be readmitted to the hospital for 2 to 3 days for a second levodopa dose-finding study, while continuing on LY300164 or placebo. After this test, patients will resume taking levodopa and the experimental drug or placebo as before for another 2 weeks.

At the end of the 2-weeks, the entire procedure will be repeated in both groups, but the treatments will be switched-that is, the patients who were taking LY300164 will now take placebo, and the patients who took placebo will now take the drug. At the end of the second 3 weeks, the levodopa infusion procedure will be repeated once more.

Throughout the study, parkinsonism symptoms and dyskinesias will be evaluated and blood samples will be drawn periodically to measure drug levels.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the acute effects of alpha-amino-3-hydroxy-5-methyl-4-isoxazole proprionic acid (AMPA) receptor blockade on the severity of parkinsonian signs and levodopa-associated motor response complications in patients with Parkinson's disease. In a controlled proof-of-principle clinical trial, efficacy will be assessed through the use of validated motor function scales. Safety will be monitored by means of frequent clinical evaluations and laboratory tests.

ELIGIBILITY:
Males and females between the ages of 30 and 75 are eligible for the study. All will carry the diagnosis of idiopathic Parkinson's disease based on the presence of a characteristic clinical history and neurological findings. All will have relatively advanced disease (Hoehn and Yahr Stages II to IV) with levodopa-associated motor response complications, including wearing-off fluctuations and peak-dose dyskinesias.

No presence or history of any medical condition that can reasonably be expected to subject the patient to unwarranted risk.

No clinically significant laboratory abnormalities including liver enzyme elevations more than three times the upper limit of normal, or neutropenia (WBC less than 4000).

No parkinson's disease patients exhibiting diphasic or end-of-dose dyskinesias or disabling dystonia.

Since LY300164 is an inhibitor of CP4503A4, patients receiving certain drugs metabolized by that pathway will not be included.

No patients who are unable to be treated with levodopa/carbidopa alone or a single, relatively short-acting dopamine agonist.

No patients who require additional treatment with amantadine or other concomitant medications.

No pregnant women or those not practicing effective means of birth control since the influence of any investigational compound on the unborn child and reproductive organs is unknown.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2000-02; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bernheimer H, Birkmayer W, Hornykiewicz O, Jellinger K, Seitelberger F. Brain dopamine and the syndromes of Parkinson and Huntington. Clinical, morphological and neurochemical correlations. J Neurol Sci. 1973 Dec;20(4):415-55. doi: 10.1016/0022-510x(73)90175-5. No abstract available. PMID 4272516
- [Background] Mizuno Y, Mori H, Kondo T. Parkinson's disease: from etiology to treatment. Intern Med. 1995 Nov;34(11):1045-54. doi: 10.2169/internalmedicine.34.1045. PMID 8774962
- [Background] Chase TN, Oh JD, Blanchet PJ. Neostriatal mechanisms in Parkinson's disease. Neurology. 1998 Aug;51(2 Suppl 2):S30-5. doi: 10.1212/wnl.51.2_suppl_2.s30. PMID 9711978